CLINICAL TRIAL: NCT01905137
Title: Botulinum Toxin Type A Versus Saline Trigger Point Injections for Myofascial Pelvic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Boston Urogynecology Associates (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Sybil Dessie, MD, Clinical Instructor, Boston Urogynecology Associates
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 015-2013
Record Dates: First submitted 2013-07-18; First posted 2013-07-23 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Myofascial Pelvic Pain
Keywords: Myofascial pelvic pain
MeSH Terms: interventions — Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botulinum Toxin Type A (Active Comparator): Patients in the treatment group will receive 200 Units of Botulinum toxin diluted in 20 mL of saline injected globally into their pelvic floor muscles followed by 8 treatments of pelvic floor physical therapy.
  Interventions: Drug: Intervention-Botulinum Toxin Type A
- Saline (Placebo Comparator): Patients in the placebo group will receive 20 mL of saline injected globally into their pelvic floor muscles followed by 8 treatments of pelvic floor physical therapy.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Intervention-Botulinum Toxin Type A — Patients will receive 200 units of Botulinum Toxin A diluted in 20 mL of preservative free saline to their pelvic floor followed by pelvic floor physical therapy.
  Other Names: Botox
  Arms: Botulinum Toxin Type A
Drug: placebo
  Other Names: saline
  Arms: Saline

SUMMARY:
The purpose of this study is to determine whether there is a change in patient-reported pelvic pain following pelvic floor injections of 200 units of Botox compared with 20cc of normal saline.

DETAILED DESCRIPTION:
Objective:

Primary objective: To evaluate the change in patient-reported pelvic pain following pelvic floor injections of 200 units of Botox compared with 20cc of normal saline.

Secondary objective: To evaluate the change in patient-reported pelvic pain following Botox injections in conjunction with pelvic floor physical therapy compared to saline injections with physical therapy.

Hypothesis We hypothesize that women in the Botox treatment arm, compared with those in the saline arm, will have a greater decrease in patient-reported pain on palpation of their most painful levator ani muscle group at two weeks after the injection.

To test this hypothesis we will measure patient-reported pain on palpation of each levator ani muscle group at baseline and two weeks following the injection. Pain will be assessed on a 10-point visual analog scale. We will compare the baseline and two-week pain measurements for the most painful muscle group.

We hypothesize that with the addition of physical therapy, women in the Botox treatment arm, compared with those in the saline arm, have a greater decrease in patient-reported pain on palpation of their most painful levator ani muscle group at 12 weeks after the injection.

To test this hypothesis we will measure patient-reported pain on palpation of each levator ani muscle group at baseline and 12 weeks following the injection. Pain will be assessed on a 10-point visual analog scale. We will compare the baseline and 12-week pain measurements for the most painful muscle group.

Intervention:

All patients will be screened for eligibility during their routine office visit. If they meet all eligibility criteria, they will be offered enrollment. At this visit, all patients will be counseled about conservative treatment options for dealing with irritative voiding symptoms, bowel symptoms, and pain. The counseling offered will be standardized for all patients. After patients are consented, they will undergo an initial evaluation with a pelvic floor physical therapist. Patients will then return for an office visit to receive their treatment. The patients will be pretreated with 100mg of topical Lidocaine hydrochloride jelly, 2%, in the vagina for 15 minutes prior to their injections. A designated medical assistant will open an opaque sealed envelope to determine whether the patient is randomized to the Botox or saline arm. The medical assistant will draw up the appropriate solution-either 20mL of saline or 200 units of Botox A diluted in preservative-free saline, to achieve a concentration of 10 units per mL. Both the Botox and saline will be drawn into 2 unlabeled 10mL syringes in order to ensure the physician remains blinded to treatment arm assignment. The saline or Botox will be injected to the coccygeus, piriformis, obturator internus, puborectalis, iliococcygeus, and pubococcygeus muscles bilaterally for a total of 1-2mL per muscle group. Using digital vaginal palpation, the muscles to be injected will be located with care taken to locate tender and contracted points on the muscle fibers. The index finger is used for palpation as the 20-gauge pudendal block needle with the guide is advanced to the target site piercing through the vaginal mucosa to the intended muscle groups. The needle is placed into the intended muscles under direct palpation for injection of 1-2mL aliquots.

Study Design:

This is a double-blinded, randomized controlled trial. Participants will be randomized to either Botox or saline in a ratio of 1:1 using computer-generated block randomization. The statistician will create the sequentially numbered opaque sealed envelopes to conceal group assignment.Study visits Baseline visit Once determined eligible, patients will be offered enrollment into the study. After consent forms are signed, we will obtain study data. Participants will then see a physical therapist at a designated pelvic floor physical therapy center to evaluate their pelvic floor prior to any intervention.

Injection visit Following the pelvic floor physical therapy assessment, participants will return to the urogynecology office for their injection of saline or Botox as specified above.

Two-week post-injection visit At two weeks, patients will return for outcome assessments. Four-week post-injection visit Patients will return at 4 weeks for the same outcome assessment they had at 2 weeks. After the 4-week visit, participants will start pelvic floor physical therapy. They will go to physical therapy for a total of 8 sessions, done as close to weekly as possible.

Twelve-week post-injection visit At 12 weeks patients will return for outcome assessments. After all outcome data are collected, the provider and the patient will be unblinded. Patients who were randomized to the placebo group will be offered 200 Units of Botox injection at no cost. These 32 patients will be encouraged to continue with weekly physical therapy for 8 weeks following the Botox injection. We will ask these participants to return at 2 weeks and 12 weeks after the injection for outcome assessments. During these visits we will collect the same data as for the 2-week and 12-week visits.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18
* Diagnosis of myofascial pain by an attending urogynecologist
* Persistent pelvic pain present for ≥50% of days over the past 3 months at a level of 6 or greater on a 10-point visual analog scale
* On physical exam, a short, tight pelvic floor with pain on palpation of at least 6 on a 10-point visual analog scale in at least one muscle group (coccygeus, pyriformis, obturator internus, iliococcygeus, puborectalis, or pubococcygeus).
* Ability to read English, provide written, informed consent and be able and willing to go to pelvic floor physical therapy.

Exclusion Criteria:

* Pregnancy or breastfeeding
* Any of the following a pre-existing neurologic or neuromuscular condition that precludes them from Botox injections, such as myasthenia gravis, a bleeding disorder; or sensitivity or allergy to Botox
* Current use of aminoglycosides or any other medication that may potentiate the neuromuscular weakness that could be caused by concomitant use of Botox also will be ineligible
* History of treatment with Botox to the pelvic floor
* Presence of any masses or lesions on physical exam
* Pelvic organ prolapse greater than stage 2
* Plan for pelvic floor surgery or pelvic floor physical therapy treatment in the next three months
* Change in pain medication usage in the past 3 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2013-07 (Actual); Primary Completion 2018-03-09 (Actual); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
To evaluate the change in patient-reported pelvic pain following pelvic floor injections of 200 units of Botox compared with 20cc of normal saline. | 2 weeks after pelvic floor injection
  To test this hypothesis we will measure patient-reported pain on palpation of each levator ani muscle group at baseline and two weeks following the injection. Pain will be assessed on a 10-point visual analog scale. We will compare the baseline and two-week pain measurements for the most painful muscle group.

SECONDARY OUTCOMES:
To evaluate the change in patient-reported pelvic pain following Botox injections in conjunction with pelvic floor physical therapy compared to saline injections with physical therapy. | 12 weeks following pelvic floor injection
  To test this we will measure patient-reported pain on palpation of each levator ani muscle group at baseline and 12 weeks following the injection. Pain will be assessed on a 10-point visual analog scale. We will compare the baseline and 12-week pain measurements for the most painful muscle group.

CONTACTS AND LOCATIONS:
Overall Officials: Eman A Elkadry, MD, Principal Investigator — Mount Auburn Hospital
Locations (1):
- Boston Urogynecology Associates, Cambridge, Massachusetts, United States

REFERENCES:
- [Derived] Dessie SG, Von Bargen E, Hacker MR, Haviland MJ, Elkadry E. A randomized, double-blind, placebo-controlled trial of onabotulinumtoxin A trigger point injections for myofascial pelvic pain. Am J Obstet Gynecol. 2019 Nov;221(5):517.e1-517.e9. doi: 10.1016/j.ajog.2019.06.044. Epub 2019 Jun 27. PMID 31254522